CLINICAL TRIAL: NCT00355017
Title: NT-BNP Guided Care in Addition to Multidisciplinary Care in Patients With Chronic Heart Failure A Three-Arm, Prospective, Randomised Study
Brief Title: BNP Guided Care in Addition to Multidisciplinary Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: VF: 05.05.2003
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2006-07

CONDITIONS: Decompensated Heart Failure

INTERVENTIONS:
Procedure: BNP-guided care in addition to multidisciplinary management

SUMMARY:
HF is associated with repeated hospitalisations and poor prognosis.The aim of this study is to investigate whether BNP-guided care (BGC) in addition to multidisciplinary management(MM) improves outcome compared to HNC alone or usual care (UC) for decompensated HF patients after discharge.

Patients hospitalised with cardiac decompensation in 9 Viennese hospitals are randomised to BGC, MM alone, or UC. MM includes 2 consultations of a heart failure (HF) specialist 10 days and 2 months after discharge for recommending medical optimisation and care by a specialised HF nurse including 4 home visits and telephone contact. In addition, BGC includes intensified increase of medical treatment during repeated follow-up visits in a HF clinic in patients with an Nt-BNP level above 2200pg/ml at discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical signs and symptoms of cardiac decompensation during the present hospitalisation
2. NYHA class III or IV at time of admission
3. Cardiothoracic ratio > 0.5, and/or left ventricular ejection fraction <40% documented by echocardiography

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-09; Study Completion 2005-09

PRIMARY OUTCOMES:
Heart failure rehospitalisation rate;
combined endpoint death or heart failure rehospitalisation;

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pacher, MD, Principal Investigator — Medical University of Vienna

REFERENCES:
- [Derived] Berger R, Moertl D, Peter S, Ahmadi R, Huelsmann M, Yamuti S, Wagner B, Pacher R. N-terminal pro-B-type natriuretic peptide-guided, intensive patient management in addition to multidisciplinary care in chronic heart failure a 3-arm, prospective, randomized pilot study. J Am Coll Cardiol. 2010 Feb 16;55(7):645-53. doi: 10.1016/j.jacc.2009.08.078. PMID 20170790